CLINICAL TRIAL: NCT00805571
Title: Urinary Kidney Injury Molecule-1 As Diagnostic Biomarker of Proximal Tubular Injury in Adult and Pediatric Transplant Recipients
Brief Title: Urinary Kidney Injury Molecule-1 (KIM-1) Excretion As Biomarker for Injury in Kidney Transplant Recipients
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Institutional Review Board, North Shore-LIJ Health System
Other Study IDs: 08-196
Record Dates: First submitted 2008-12-05; First posted 2008-12-09 (Estimated); Last update posted 2010-03-12 (Estimated); Status verified 2010-03

CONDITIONS: Kidney Transplant Dysfunction
Keywords: Rejection; Infection; Side effect of immunosuppressive drug (nephrotoxicity)
MeSH Terms: conditions — Rejection, Psychology; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Adult: Adult patients with end-stage kidney disease awaiting kidney transplantation.
- Pediatric: Children with end-stage kidney disease awaiting kidney transplantation.

SUMMARY:
The purpose of this study is to determine if measuring the level of a protein called Kidney Injury Molecule-1 (KIM-1) in the urine will help healthcare providers detect any problems with the transplanted kidney before the laboratory investigations that are used on a routine basis do. This approach may allow the doctor to intervene at an earlier point of a rejection episode and may thereby prolong survival of the transplant kidney.

DETAILED DESCRIPTION:
SPECIFIC AIMS:

1. To investigate the role of urinary Kim-1 excretion as a marker of delayed graft function, acute kidney allograft rejection and/or virus-induced allograft nephropathy and/or calcineurin-inhibitor nephrotoxicity.
2. To determine the role of urinary Kim-1 excretion in predicting long term outcome after kidney transplantation compared to standard diagnostic tests.
3. To determine the role of reduction in urinary Kim-1 excretion after a rejection episode and/or viral infection as a marker of repair of renal tubules.

HYPOTHESIS:

Monitoring of urinary KIM-1 in kidney transplant recipients will facilitate the detection of delayed graft function, acute allograft rejection or infectious causes of proximal tubular injury, allowing earlier intervention with better long-term graft survival. Detection of urinary KIM-1 will precede increases in serum creatinine to detect acute graft injury and urinary KIM-1 will decrease faster than serum creatinine and will predict responsiveness (or lack thereof) to intervention more accurately.

ELIGIBILITY:
Inclusion Criteria:

Children and adults from the age of 3 years who are eligible transplant candidates listed for deceased donor kidney or who are scheduled for a living related or unrelated donor kidney transplant at Mount Sinai Hospital will be eligible for inclusion in this project. Patients will be recruited from the population awaiting kidney transplant treated at the Schneider Children's Hospital and Mount Sinai Hospital.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adult and pediatric patients with chronic renal failure who are listed at Mount Sinai Hospital for a deceased donor kidney transplant and/or who are in the process of having a living donor evaluation are eligible to participate. One urine sample will be sent for KIM-1 measurement before transplantation, once the patient or the caregiver of the patient consents to participation in the study. The next specimen of urine will only be collected status post kidney transplant in the immediate post-operative phase and on routine visits thereafter. The study does not require obtaining any extra blood or urine specimens, but uses urine that would otherwise be discarded.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2008-10; Primary Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice Goilav, MD, Principal Investigator — Northwell Health
Locations (1):
- Schneider Children's Hospital, New Hyde Park, New York, United States